CLINICAL TRIAL: NCT05104138
Title: OCTA in Central Serous Chorioratinopathy Treated With Oral Eplerenone or Hal-fluence Photodynamic Therapy: a Comparative Study
Brief Title: Eplerenone Versus PDT: Comparative Study by OCTA
Status: Completed | Type: Observational
Sponsor: Federico II University (Other)
Responsible Party: Principal Investigator, Gilda Cennamo, Principal Investigator, Federico II University
Other Study IDs: 1010/2021
Record Dates: First submitted 2021-10-21; First posted 2021-11-02 (Actual); Last update posted 2021-11-02 (Actual); Status verified 2021-10

CONDITIONS: Central Serous Chorioretinopathy
MeSH Terms: conditions — Central Serous Chorioretinopathy | interventions — Eplerenone; Dosage Forms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Half fluence photodynamic therapy: Patients with central serous chorioretinopathy, treated by half-fluence photodynamic therapy
  Interventions: Device: The patients underwent half fluence photodynamic therapy for 6 months
- Oral Eplerenone: Patients with central serous chorioretinopathy, treated by oral eplerenone
  Interventions: Drug: Eplerenone

INTERVENTIONS:
Drug: Eplerenone — The patients underwent eplerenone treatment for 6 months
  Other Names: Eplerenone in oral dose form
  Groups: Oral Eplerenone
Device: The patients underwent half fluence photodynamic therapy for 6 months — Half fluence photodynamic therapy for 6 months
  Groups: Half fluence photodynamic therapy

SUMMARY:
The study aims to analyze the changes in OCTA parameters and in choroidal thickness in patients affected by central serous chorioretinopathy treated by oral eplerenone and half-fluence photodynamic therapy.

DETAILED DESCRIPTION:
Central serous chorioretinopathy (CSC) is a chorioretinal disease characterized by serous detachment due to the dilatation and hyperpermeability of choroidal vessels resulting in the accumulation of serous fluid between the neurosensory retina and the retinal pigment epithelium.

Several studies reported the efficacy of half-fluence photodynamic therapy (PDT) and oral eplerenone in the CSC treatment inducing a reduction of the choroidal hyperpermeability and remodeling the choroidal vascularization.

This retrospective study aims to perform a quantitative analysis of retinal and CC vessel density by OCTA at baseline, 3 and 6 months in patients underwent PDT and patients underwent eplerenone.

ELIGIBILITY:
Inclusion Criteria:

* age older than 30 years
* diagnosis of central serous chorioretinopathy
* treatment-naïve with half-fluence photodynamic therapy or oral eplerenone
* absence of vitreoretinal and vascular retinal diseases

Exclusion Criteria:

* age younger than 30 years
* absence of diagnosis of central serous chorioretinopathy
* previous treatment with half-fluence photodynamic therapy or oral eplerenone
* presence of concomitant vitreoretinal and vascular retinal diseases

Ages: 30 Years to 60 Years | Sex: All
Age Groups: Adult
Study Population: The participans were older than 40 years with central serous chorioretinopathy. They did not present other ophthalmological diseases
Sampling Method: Non-Probability Sample
Enrollment: 30 (Actual)
Dates: Start 2015-10-01 (Actual); Primary Completion 2017-10-30 (Actual); Study Completion 2017-11-30 (Actual)

PRIMARY OUTCOMES:
Study of vessel density in retinal choriocapillaris networks, using OCTA, in patients underwent half fluence photodynamic therapy and oral eplerenone | 6 months
  To evaluate the role of optical coherence tomography angiography in predicting the changes of the vessel density of retinal and choriocapillaris vascular networks , comparing patients underwent half-fluence phodynamic therapy and patients with oral eplerenone.
  The vessel density are expressed as percentage

CONTACTS AND LOCATIONS:
Overall Officials: Gilda Cennamo, Principal Investigator — Università Federico II